CLINICAL TRIAL: NCT05520060
Title: The Effect of Continuous Midwifery Care at Birth on Labor Pain, Comfort and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ayseren Cevik, Lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03.06.2022/49
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Labor Pain
Keywords: Continuous midwifery care; supportive care; Labor pain; Comfort,
MeSH Terms: conditions — Labor Pain | interventions — Palliative Care; Environment; Delivery of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): The experimental group will be placed in continuous midwifery care. The continuous and supportive care stages to be presented at birth are planned within the framework of Kolcaba's comfort theory. According to this theory, interventions will be applied according to the physical, psychospiritual, environmental and sociocultural comfort needs of women.
  Interventions: Other: Physical support; Other: Psychospiritual support; Other: Environmental and sociocultural support; Other: Routine care
- Control (Placebo Comparator): The experimental group will be placed in routine midwifery care.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Physical support — Pharmacological and non-pharmacological methods in pain management, Mobilization, Position preferred by the woman, Fluid and nutritional support, Massage applications, Sacral pressure, Listening to music, Breathing and relaxation exercises
  Other Names: Supportive Care
  Arms: experimental
Other: Psychospiritual support — Effective communication, Encouragement to speak up and express fears, Support for faith-oriented practices
  Other Names: Supportive Care
  Arms: experimental
Other: Environmental and sociocultural support — egulating the temperature, light and sound of the room, Environment that promotes respect for privacy, Reducing environmental noise, Information, Social support, Talking about cultural practices, Social support
  Other Names: Supportive Care
  Arms: experimental
Other: Routine care — Admission to the delivery room, preparation for birth, delivery, postpartum care, etc.
  Other Names: Health care

SUMMARY:
Introduction: Birth is a period in which biological, physical, emotional and social changes are experienced. Supportive care provided by the midwife ensures the adaptation of the woman to labor and improves her ability to cope with labor. Supportive care has positive effects on labor and maternal and infant health.

Purpose: This project aimed to determine the birth pain, comfort and satisfaction levels by considering the continuous midwifery care at birth with a holistic approach.

Method: The universe of this study, which will be conducted in randomized controlled experimental type, will consist of pregnant women who applied to Adana City Training and Research Hospital, Gynecology and Obstetrics Clinic, Delivery Room. The number of samples was calculated by G*power analysis, and it was aimed to carry out the research with 30 participants in the intervention group and 30 participants in the control group. Single-blind randomized assignment and block randomization will be performed to avoid selection bias. Data will be collected using face-to-face interview technique. The pre-test will be applied to pregnant women who apply to the delivery room in the latent phase. While the continuous midwifery care model will be applied to the intervention group, standard midwifery care will be applied to the control group. The final test will be done between 1-4 hours postpartum. The independent variable of the study is continuous midwifery care. The dependent variable is the introductory characteristics of women, labor pain, comfort and satisfaction levels. The data will be analyzed with appropriate analysis methods after performing normality tests.

DETAILED DESCRIPTION:
During childbirth, women need someone's support. Providing continuous care to women with a supportive and holistic approach by midwives who care for women is seen as a potential that can improve labor pain management, birth comfort and satisfaction. The aim of this research is to determine the effect of continuous midwifery care at birth on labor pain, comfort and satisfaction levels.

For this purpose, the objectives are:

* To apply the continuous midwifery care model,
* To increase women's normal birth comfort and satisfaction,
* To create social awareness that midwives play a key role in normal birth,
* Reducing preventable maternal and infant and infant deaths due to care deficiencies,
* To reduce cesarean rates.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate
* Knowing Turkish and being literate,
* Don't be in the latent phase.

Exclusion Criteria:

* high risk pregnancy
* Multiple pregnancy
* Breech presentation
* Induction of labor
* Emergency cesarean section indication

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants are women who have given birth.
Enrollment: 60 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Birth Comfort Scale | pre-intervention/passive phase of childbirth; immediately after the intervention/active phase of childbirth. An increase in the score is interpreted as an increase in comfort level.
  Change from birth comfort between passive phase of childbirth and active phase of childbirth.
Birth Satisfaction Scale | immediately after the intervention/1-4 hours postpartum. An increase in the score is interpreted as an increase in satisfaction level.
  Birth satisfaction in the early postpartum period.
Scale of Pain Expression during Childbirth (ESVADOPA) | pre-intervention/passive phase of childbirth; immediately after the intervention/active phase of childbirth.An increase in the score is interpreted as an increase in the expression of pain.
  Change from pain expression level between passive phase of childbirth and active phase. of childbirth.
Visual Analog Scale | pre-intervention/passive phase of childbirth; immediately after the intervention/active phase of childbirth. An increase in the score is interpreted as an increase in pain.
  Change from pain between passive phase of childbirth and active phase of childbirth.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No